CLINICAL TRIAL: NCT05804201
Title: A Prospective, Single-center, Single-arm Study to Evaluate the Safety and Effectiveness of a Long Partially Covered Metal Stent With Hot Delivery System (Hot Giobor) for EUS-guided HGS in Patients With Malignant Biliary Obstruction
Brief Title: EUS-guided Hepatico-gastrostomy With Hot Giobor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN SHANNON MELISSA, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022.460
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Malignant Biliary Obstruction
Keywords: EUS-guided hepatico-gastrostomy, malignant biliary obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HOT Giobor (Other): EUS-guided hepatico-gastrostomy would be performed with Niti-S HOT Giobor (Taewoong Medical, Gyeonggi-do, Korea), a novel device designed for hepatico-gastrostomy.
  Interventions: Procedure: EUS-guided hepatico-gastrostomy would be performed with Niti-S HOT Giob

INTERVENTIONS:
Procedure: EUS-guided hepatico-gastrostomy would be performed with Niti-S HOT Giob — (2) The EUS procedure will be performed with a therapeutic echoendoscope with a large working channel under guidance of ultrasound, endoscopy, and fluoroscopy. The echoendoscope will be positioned in the stomach or duodenum. Liver segment III, or sometimes segment II, will be punctured with an 19G needle. After puncture, a guidewire will be introduced in the dilated bile duct, and a Hot Giobor will be placed. All procedures will be performed with the patient and in the supine or prone position under monitored anesthesia.

SUMMARY:
Endoscopic ultrasonography-guided hepaticogastrostomy (EUS-HGS) is a method of obtaining biliary drainage in patients with failed or difficult endoscopic retrograde cholangiopancreatography (ERCP). The reason for failure of ERCP can be due to gastric outlet obstruction or failed cannulation. HGS involves placement of a stent between the bile duct and the stomach under the guidance of endoscopic ultrasound to create a biliary drainage route similar to surgery. The overall reported success rate is 94% with an overall complication rate of 14%. The most common complications include pneumoperitoneum (air leaking into the abdomen) and bile leak. Both complications are usually managed conservatively. EUS-gudied HGS has been commonly performed but the type of stent used for the procedure is still under evolution. A specific stent is needed to prevent complications. The most commonly used stent in HK is a hybrid stent where the liver portion is uncovered to avoid stent migration and the rest of the stent is covered to avoid bile leakage and pneumoperitonum. This stent is already available and is called the Giobor stent. However, in order to use this stent, during the EUS procedure, the bile duct needs to be first punctured by a EUS needle, then a guidewire passed, then dilate the tract with an energy deviced 6Fr cytotome, then the stent can be passed. This process is cumbersome and increase the chance of complications during exchange of the devices. A newly developed stent that is cautery-fitted has been developed. The use of this stent shortens the steps of stent application. The current study aims to evaluate the feasibility and safety of a novel stent that is cautery-fitted designed for performance of EUS-HGS (Niti-S HOT Giobor).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients ≥ 18 years old
* Anatomically feasible for EUS-guided hepatico-gastrotomy
* Patient with clinical symptoms and/or sign of extra-hepatic biliary obstruction (jaundice, biliary-type pain, cholangitis)
* Patients with unsuccessful ERCP (failed ECRP, anticipated difficult ERCP or high risk for pancreatitis)
* Written informed consent (and assent when applicable) obtained from subject

Exclusion Criteria:

* Severe comorbidities precluding the endoscopic procedure (such as cardiopulmonary disease, sepsis, or a bleeding disorder)
* Life expectancy of less than 1 month
* History of gastric surgery
* Coagulation disorders
* Pregnancy, breastfeeding, or unwilling to practice birth control during participation in the study
* Severe allergy to Nickel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedural / Device related serious adverse events | 1 month
  Any related serious adverse events occured in 1 month post procedure
Bilirubin level improvement | 1 month
  Bilirubin level improvement is defined as: > 50% serum bilirubin level is decreased from baseline.

SECONDARY OUTCOMES:
Technical success | During index procedure
  Hot Giobor stent is placed at the desired site: transmural placement of the Hot Giobor stent across the stomach or duodenum into the bile duct.
Clinical success | At day 7
  Bilirubin level improvement is defined as: >20% serum bilirubin level is decreased from baseline.
Stent patency | At 3, 6, 9 and 12 months
  Time between stent placement and stent occlusion &/or stent removal.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Melissa Chan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese Universtiy of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No